CLINICAL TRIAL: NCT03375918
Title: COmmuNity-engaged SimULation Training for Blood Pressure Control
Acronym: CONSULT-BP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Jennifer Tjia, Professor of Population and Quantitative Health Sciences, University of Massachusetts, Worcester
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: H00012160; 1R01MD011532 (NIH)
Record Dates: First submitted 2017-12-12; First posted 2017-12-18 (Actual); Results first posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-08

CONDITIONS: Hypertension
Keywords: Healthcare disparities; Racial Bias
MeSH Terms: conditions — Hypertension; Racism

STUDY DESIGN:
Intervention Model Description: Enrolled 4 sequential cohorts of clinical trainees [stratified by specialty (internal medicine (IM), family medicine (FM)] were to be assigned to 1 of 5 start dates within each cohort year. During the global pandemic, randomized assignment within each year was not possible due to clinical needs of the hospitals, which means that the intervention was a pre-post intervention study. Clinical outcomes will be assessed at the patient level.
Masking Description: The primary outcome is blood pressure (BP) change as recorded in the electronic medical record (EMR) of racial/ethnic minority patients and Medicaid recipients of any race/ethnicity with controlled and uncontrolled hypertension. Secondary outcomes are standardized patient assessments of clinical trainee communication skills. Standardized patient participants are masked to the intervention status of their provider trainees.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthcare Trainees (Other): Trainees were assigned to receive Other: CONSULT-BP Educational Intervention. Each arm has a pre-intervention (control) period and a post-intervention (exposure) period.
  Interventions: Other: CONSULT-BP Educational Intervention

INTERVENTIONS:
Other: CONSULT-BP Educational Intervention — CONSULT-BP is a two sessions training provided to healthcare trainees over a 5-week period. The first session focused on (1) didactic overview of healthcare disparities, social drivers of health, implicit bias and systemic racism and (2) interactive discussions and patient storytelling videos to raise awareness of the bi-directional role of racial and ethnic identity among clinicians and patients. The second session focused on skill building and included (1) bias mitigation strategies based on the RELATE bias mitigation tool and (2) skill practice using 2 standardized patient simulated clinical encounters focusing on hypertension management challenges.

SUMMARY:
The goal of CONSULT-BP is to train early-stage healthcare providers, including residents and nurse practitioner (NP) students, to mitigate providers' bias, improve communication skills, and enhance providers' ability to develop authentic and meaningful therapeutic alliances with patients. The study setting is an academic safety net hospital that serves a large non-White and poor population. The Investigators hypothesize that patients' outcomes (blood pressure levels) will be lower after the training intervention compared with before training (control) periods.

DETAILED DESCRIPTION:
CONSULT-BP is an intervention to test a theory-based, 'awareness, exposure and skill-building' approach applied in the safety of a simulation-based learning center, to improve providers' interaction skills with minority and poor patients. The study included community-based participatory research input to develop and implement CONSULT-BP in an academic medical center with a large, safety-net health system which serves minority and poor population.

ELIGIBILITY:
For Healthcare Trainees -

Inclusion Criteria:

1. Practice at a clinical site supported by an EMR to allow clinical data collection for outcome measurement
2. 15-week clinical look-back period
3. No prior completion of the CONSULT-BP intervention

Exclusion Criteria: 1. All 1st year trainees

For Patient Participants -

Inclusion Criteria:

1. English-speaking
2. Non-White racial/ethnic minority or Medicaid recipient (regardless of race/ethnicity)
3. Hypertension identified in the EMR

Exclusion Criteria:

1. Enrolled in hospice.
2. Pregnancy, dementia, schizophrenia, bipolar illness, or other serious medical co-morbidity that would interfere with hypertension self-control

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2024-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Tjia, MD, MSCE, Principal Investigator — UMass Medical School
Locations (4):
- United States (4):
  - Barre Family Health Center, Barre, Massachusetts
  - Tri River Family Health Center, Uxbridge, Massachusetts
  - UMass Memorial Hahnemann Family Health Center, Worcester, Massachusetts
  - UMass Memorial Medical Center -- Benedict Building, Worcester, Massachusetts

IPD SHARING:
Plan to Share IPD: No
Individual level participant data includes protected health information. There is no plan to share these data with other researchers.

REFERENCES:
- [Background] Tjia J, Pugnaire M, Calista J, Eisdorfer E, Hale J, Terrien J, Valdman O, Potts S, Garcia M, Yazdani M, Puerto G, Okero M, Duodu V, Sabin J. Using Simulation-Based Learning with Standardized Patients (SP) in an Implicit Bias Mitigation Clinician Training Program. J Med Educ Curric Dev. 2023 Jun 5;10:23821205231175033. doi: 10.1177/23821205231175033. eCollection 2023 Jan-Dec. PMID 37324051
- [Background] Tjia J, Pugnaire M, Calista J, Esparza N, Valdman O, Garcia M, Yazdani M, Hale J, Terrien J, Eisdorfer E, Zolezzi-Wyndham V, Chiriboga G, Rappaport L, Puerto G, Dykhouse E, Potts S, Sifuentes AF, Stanhope S, Allison J, Duodo V, Sabin J. COmmuNity-engaged SimULation Training for Blood Pressure Control (CONSULT-BP): A study protocol. Medicine (Baltimore). 2021 Feb 5;100(5):e23680. doi: 10.1097/MD.0000000000023680. PMID 33592827
- [Background] Calista J, Esparza N, Fernandez J, Beltran A, Bradshaw J, Casseres A, Duodu S, Duodu V, Fordjour C, Kuffour B, Mensah L, Negron-Cruz L, Pietri C, Pridgen C, Puerto G, Tessler LA, Tucci S, Wood K, Wright S, Zinkus P, Tjia J. Perspectives of Community Partners Involved in an Academic Training to Address Clinicians' Implicit Bias. Prog Community Health Partnersh. 2023;17(2):347-351. doi: 10.1353/cpr.2023.a900215. PMID 37462563

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Within each academic year, we aimed to randomize training times to 1 of 5 start dates using a stepped wedge design. However, this design was not feasible beyond the first year of our study because of the COVID emergency.
Pre-assignment Details: To maintain clinical staff services in the hospital, we were not able to maintain the cluster randomization of trainees. We aimed to enroll cohorts of trainees over a 3-year period, with each academic year constituting an intervention cycle, with 3 cycles of implementation corresponding to 3 sequential academic years. Due to COVID, we extended enrollment to a 4-year period.
  Please note - only trainee participants were considered enrolled. Patient participants were not considered 'enrolled'.
Groups:
- Year 1: Start Time 1: 1 of 5 trainee groups to start the intervention at time point 1.
- Year 1: Start Time 2: 1 of 5 trainee groups to start the intervention at time point 2.
- Year 1: Start Time 3: 1 of 5 trainee groups to start the intervention at time point 3.
- Year 1: Start Time 4: 1 of 5 trainee groups to start the intervention at time point 4.
- Year 1: Start Time 5: 1 of 5 trainee groups to start the intervention at time point 5.
- Year 2: Cohort 1: Trainees in year 2
  Outcomes measured at level of patients nested within trainee Control period patient BP measures are pre-intervention Intervention period patient BP measures are post-intervention
- Year 3: Cohort 2: Trainees in year 3
  Outcomes measured at level of patients nested within trainee Control period patient BP measures are pre-intervention Intervention period patient BP measures are post-intervention
- Year 4: Cohort 3: Trainees in year 4
  Outcomes measured at level of patients nested within trainee Control period patient BP measures are pre-intervention Intervention period patient BP measures are post-intervention
Period: Overall Study
Arm/Group | Year 1: Start Time 1 | Year 1: Start Time 2 | Year 1: Start Time 3 | Year 1: Start Time 4 | Year 1: Start Time 5 | Year 2: Cohort 1 | Year 3: Cohort 2 | Year 4: Cohort 3
Started | 600 | 106 | 527 | 215 | 264 | 336 | 256 | 409
Control Patients (Control Period Measurements for Patients Nested within Trainee before the Intervention Training) | 54 | 40 | 201 | 104 | 125 | 150 | 80 | 190
Intervention Patients (Intervention Period Measurements for Patients Nested within Trainee Post-Intervention Training) | 534 | 60 | 314 | 98 | 135 | 159 | 155 | 196
Trainees (Trainees Completing Intervention Outcomes measured at level of patients nested within trainee The same trainee participants participated in, and treated patients, in both the Control and Intervention periods of the study.) | 12 | 6 | 12 | 13 | 4 | 27 | 21 | 23
Completed | 600 | 106 | 527 | 215 | 264 | 336 | 256 | 409
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline information on Healthcare Trainees, Patients--Control Arm and Patients--Intervention Arm are aggregated from all cohorts within each population.
Groups:
- Healthcare Trainees: Healthcare trainee clusters assigned to 1 of 5 start dates training times for Other: CONSULT-BP Educational Intervention. Each arm has a pre-intervention (control) period and a post-intervention (exposure) period.
- Patients - Control Arm: Patients treated by healthcare trainees within the control period
- Patients - Intervention Arm: Patients treated by healthcare trainees within the intervention period
- Total: Total of all reporting groups
Arm/Group | Healthcare Trainees | Patients - Control Arm | Patients - Intervention Arm | Total
Number analyzed (Participants) | 118 | 944 | 1651 | 2713
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.7 (2.75) | 54.8 (13.6) | 54.8 (13.2) | 54.8 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 486 | 894 | 1438
  Male | 60 | 458 | 757 | 1275
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 135 | 217 | 361
  Not Hispanic or Latino | 53 | 800 | 1425 | 2278
  Unknown or Not Reported | 56 | 9 | 9 | 74
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 22 | 81 | 117 | 220
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 214 | 364 | 582
  White | 39 | 215 | 383 | 637
  More than one race | 1 | 425 | 778 | 1204
  Unknown or Not Reported | 52 | 9 | 9 | 70
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 118 | 944 | 1651 | 2713

OUTCOME MEASURES:

1. Primary Outcome: Blood Pressure
Description: Systolic and diastolic blood pressure of patients treated by the participating clinician trainees as reported in the Electronic Medical Record.
Time Frame: Control period is 6 months before the intervention and intervention period is up to 6 months after the intervention
Population: Blood pressure data was obtained from electronic medical records of 944 patients during the control period and 1,651 period patients during the intervention period.
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- Patients - Pre CONSULT-BP Intervention: Patient BPs from prior to the CONSULT-BP Intervention taken from the Electronic Medical Record.
- Patients - Post-Intervention: Patient BPs from after the CONSULT-BP Intervention taken from the Electronic Medical Record.
Arm/Group | Patients - Pre CONSULT-BP Intervention | Patients - Post-Intervention
Number analyzed (Participants) | 944 | 1651
mm Hg
  Systolic Blood Pressure | 137.6 (18.6) | 136.4 (18.6)
  Diastolic BloodPressure | 82.1 (11.1) | 81.8 (10.8)

2. Secondary Outcome: RELATE Checklist, a Standardized Patient Rating Scale for Bias-Mitigating and Patient-Centered Communication
Description: The RELATE (Respect, Empathize, Listen, Ask, Talk, Engage) is a 19-item checklist completed by an informant group of "standardized" patients during a simulated standardized patient encounter to evaluate interaction with the participating clinicians. The RELATE checklist contains 4 factors: Respect (4 items), Empathetic Listening (5 items); Ask and Talk (Inquiry, 6 items), and Engagement in Partnership (4 items). The checklist scores are from 0 to 38, with higher scores reflecting better communication from the perspective of the "standardized" patient.
Time Frame: During CONSULT-BP session 2 clinician training intervention (simulated standardized patient encounter)
Population: RELATE scores were obtained from "standardized patients" (or mock patients) during interaction with the Clinician Trainees.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Healthcare Trainees: Within each academic year, trainee clusters are assigned1 of 5 start date training times for Other: CONSULT-BP Educational Intervention. Each arm has a pre-intervention (control) period and a post-intervention (exposure) period.
  CONSULT-BP Educational Intervention: Our intervention comprised two sessions over a 5-week period. The first session focused on (1) didactic overview of healthcare disparities, social drivers of health, implicit bias and systemic racism and (2) interactive discussions and patient storytelling videos to raise awareness of the bi-directional role of racial and ethnic identity among clinicians and patients. The second session focused on skill building and included (1) bias mitigation strategies based on the RELATE bias mitigation tool proposed by Cooper (Cooper L. Why Are Health Disparities Everyone's Problem? . Baltimore: Johns Hopkins University Press; 2021.) and (2) skill practice using 2 standardized patient simulated clinical encounters focusing on hypertension management challenges. The second session lasted 4 hours. Between the two sessions, trainees were asked to complete a race/ethnicity-compliance implicit association test and were provided the results to build self-awareness of potential implicit bias.
Arm/Group | Healthcare Trainees
Number analyzed (Participants) | 118
score on a scale | 32.7 (5.0)

ADVERSE EVENTS:
Time Frame: 6 months after the intervention
Description: No adverse events (defined as "Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research") were expected or noted among the participating healthcare trainees who received this educational intervention Patients did not have adverse events collected.
Groups:
- Patients - Control Arm: Patients clustered within trainees in pre-training control period
- Patients - Intervention Arm: Patients clustered within trainees in post-training intervention period
Arm/Group | Healthcare Trainees | Patients - Control Arm | Patients - Intervention Arm
All-Cause Mortality (participants affected / at risk) | 0/118 | 0/944 | 0/1651
Serious Adverse Events (participants affected / at risk) | 0/118 | 0/944 | 0/1651
Other Adverse Events (participants affected / at risk) | 0/118 | 0/944 | 0/1651

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-20): https://cdn.clinicaltrials.gov/large-docs/18/NCT03375918/Prot_SAP_000.pdf